CLINICAL TRIAL: NCT06735313
Title: Evaluation of Salivary Asprosin, IL-39,IL-40 and IL-1β Levels in Diabetic Patients with Periodontitis
Brief Title: Changes in Salivary Asprosin, IL-39, IL-40 and IL-1β Levels in Diabetic Patients with Periodontitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, AYSE HUMEYRA ORUC, research assistant, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: periodontitisanddiabetes
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus; Periodontal Disease; Asprosin; Interleukin 1-beta
MeSH Terms: conditions — Diabetes Mellitus; Periodontal Diseases; Arachnodactyly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Periodontally healthy, systemically healthy individual (Other): Before starting the treatment of the patients and after each planned treatment, routine periodontal status records (periodontal pocket depths of the teeth, attachment losses, mobility levels, furcation defect degrees, bleeding index on probing, gingival index, plaque index, amount of keratinized gingiva, gingival recession, body/mass index) are taken and archived. In addition, sociodemographic data and brushing habits of each patient participating in the study are recorded. Saliva samples will also be collected from the patients before the treatment.
  Interventions: Diagnostic Test: Periodontal examination and saliva collection
- periodontally healthy individuals with type 2 diabetes (Active Comparator): Before starting the treatment of the patients and after each planned treatment, routine periodontal status records (periodontal pocket depths of the teeth, attachment losses, mobility levels, furcation defect degrees, bleeding index on probing, gingival index, plaque index, amount of keratinized gingiva, gingival recession, body/mass index) are taken and archived. In addition, sociodemographic data and brushing habits of each patient participating in the study are recorded. Saliva samples will also be collected from the patients before the treatment.
  Interventions: Diagnostic Test: Periodontal examination and saliva collection
- Systemically healthy individual with periodontitis (Active Comparator): Before starting the treatment of the patients and after each planned treatment, routine periodontal status records (periodontal pocket depths of the teeth, attachment losses, mobility levels, furcation defect degrees, bleeding index on probing, gingival index, plaque index, amount of keratinized gingiva, gingival recession, body/mass index) are taken and archived. In addition, sociodemographic data and brushing habits of each patient participating in the study are recorded. Saliva samples will also be collected from the patients before the treatment.
  Interventions: Diagnostic Test: Periodontal examination and saliva collection
- Individual with periodontitis and type 2 diabetes (Active Comparator): Before starting the treatment of the patients and after each planned treatment, routine periodontal status records (periodontal pocket depths of the teeth, attachment losses, mobility levels, furcation defect degrees, bleeding index on probing, gingival index, plaque index, amount of keratinized gingiva, gingival recession, body/mass index) are taken and archived. In addition, sociodemographic data and brushing habits of each patient participating in the study are recorded. Saliva samples will also be collected from the patients before the treatment.
  Interventions: Diagnostic Test: Periodontal examination and saliva collection

INTERVENTIONS:
Diagnostic Test: Periodontal examination and saliva collection — Before the periodontal examination, saliva samples are collected from each patient participating in the study and periodontal measurements are made.

SUMMARY:
The aim of this study is to determine the relationships between asprosin, IL-39, IL-40 and IL-1β in saliva between individuals with and without diabetes and between individuals with periodontitis and healthy individuals and to determine the potential roles of these biomarkers that are multiplied in periodontal disease. The study aims to evaluate whether these biomarkers can be used for periodontal diagnosis or prognosis.

The questions answered by the study are as follows:

Do asprosin, IL-39, IL-40 and IL-1β biomarker levels differ between individuals with and without diabetes? Do these biomarker levels differ significantly between individuals with periodontitis and individuals who are healthy? Can these biomarkers be used in the early diagnosis or recording the progression of periodontal diseases?

DETAILED DESCRIPTION:
The study is planned to be conducted with 176 individuals with and without periodontal disease between the ages of 18-80 who come to the Department of Periodontics of the Faculty of Dentistry of Necmettin Erbakan University for treatment. Those who sign the 'informed consent form' will be included in the study.

In the periodontal examination of each patient who applies to the periodontology clinic, routine radiographic and clinical evaluations are performed, and routine periodontal status records (periodontal pocket depths of the teeth, attachment losses, mobility levels, furcation defect degrees, bleeding index on probing, gingival index, plaque index, amount of keratinized gingiva, gingival recessions, body/mass index) are taken and archived before the start of the patients' treatments and after each planned treatment. In addition, the sociodemographic data and brushing habits of each patient who will participate in the study are recorded. Saliva samples will also be collected from patients prior to treatment. Individuals will be divided into groups according to their periodontal disease status:

* 44 periodontally healthy, systemically healthy individuals
* 44 periodontally healthy, type 2 diabetic individuals
* 44 periodontitis, systemically healthy individuals
* 44 periodontitis, type 2 diabetic individuals

A calibrated expert clinician will determine periodontal status according to the criteria of the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions based on radiographic and clinical examination. Patients will need to meet the criteria for Stage II and III, generalized, periodontitis to be included in the periodontitis groups.

Saliva samples will be collected before periodontal measurements are taken to prevent saliva from bleeding during probing. Participants will be asked not to brush their teeth at least one hour before the sample collection and to avoid any food, sugary gum, cosmetic products such as lipstick, and any medication that will not affect the salivary hormone measurements. A total of 5 2 ml samples, one for each marker, will be collected from each patient between 9:00 and 10:00 in the morning. The samples will be collected in plastic tubes with a glass funnel within five minutes after each participant rinses their mouth with water. The tubes will then be capped and the samples will be centrifuged at 1000 rpm for 10 minutes to remove cellular elements and plaque. The supernatant liquid will be pipetted without touching the sediment formed at the bottom of the tubes, placed in polypropylene Eppendorf tubes, and stored at -20°C until analysis.

Analysis of Saliva Samples Samples will be placed at +4°C to be thawed on the day of analysis. ELISA kits will be used to determine Asprosin, IL-39,IL-40, IL-38 and IL-1B levels according to the manufacturer's instructions (Elabscience Biotechnology Co. Ltd).

Statistical Analysis Statistical analysis will be performed using the Statistical Package for Social Sciences (SPSS) version 23 (IBM Corp., Armonk, NY).

Data will be expressed as mean and standard deviation. Data normality will be assessed using the Kolmogorov-Smirnov test. Differences between parameter means in intragroup comparisons of periodontally healthy and periodontitis groups will be assessed using the One-way ANOVA (Bonferroni post-hoc) test. Differences between parameter means between periodontally healthy and periodontitis groups will be assessed using the independent t test. Pearson correlation coefficients will be used to assess correlations between clinical and biochemical parameters. Areas under the curve (AUC) and receiver operating characteristic (ROC) curves will be used to examine the sensitivity and specificity of salivary biomarkers in distinguishing periodontitis from periodontal health. p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:- No systemic disease such as nephrotic syndrome, chronic renal disease and cardiovascular disease

* No dental scaling and root planing treatment in the last 6 months
* No antibiotic use for any reason
* Having at least 20 teeth in the mouth
* Not being pregnant or breastfeeding

Inclusion criteria for the periodontally healthy group

* Having a periodontally healthy diagnosis in routine clinical and radiographic examinations Inclusion criteria for the periodontitis group
* Diagnosing periodontitis in routine clinical and radiographic examinations

Exclusion Criteria:

* - Patients with any autoimmune disease (Rheumatoid arthritis, familial Mediterranean fever, ankylosing spondylitis, Behcet, psoriasis, etc.) - Those who smoke 10 or more cigarettes per day

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
measurement of preoperative periodontal parameters | before collecting saliva
  To determine the baseline condition, preoperative measurement of periodontal parameters (amount of keratinized tissue, papilla height, papilla width, probing pocket depth, amount of recession, tissue thickness) will be recorded in millimeters using a periodontal probe.
gingival index measurement | before collecting saliva
  The status of gingival health will be assessed using the Gingival Index (Loe and Silness, 1963). This measurement will be made to determine the degree of gingival inflammation and will be scored on a scale from 0 (healthy gingiva) to 3 (severe inflammation and bleeding).
  Unit of Measurement: 0-3 scale.
Plaque Index (PI) measurement | before collecting saliva
  The degree of plaque accumulation on the tooth surfaces will be assessed using the Plaque Index (Silness and Loe, 1964). The assessment will be made on a scale from 0 (no plaque) to 3 (entire tooth surface covered with plaque). This measurement will be used to objectively determine the degree of plaque formation.Unit of Measurement: 0-3 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

REFERENCES:
- [Background] Gul SNS, Eminoglu DO, Laloglu E, Aydin T, Dilsiz A. Salivary and serum asprosin hormone levels in the 2018 EFP/AAP classification of periodontitis stages and body mass index status: a case-control study. Clin Oral Investig. 2024 Jan 13;28(1):91. doi: 10.1007/s00784-024-05494-9. PMID 38217801
- [Derived] Oruc AH, Babayigit O. Salivary asprosin, IL-39, IL-40, and IL-1beta levels in diabetic patients with periodontitis: A cross-sectional analysis. Clin Oral Investig. 2026 Jan 14;30(1):52. doi: 10.1007/s00784-026-06744-8. PMID 41530539